CLINICAL TRIAL: NCT03118076
Title: The Effect of Dexmedetomidine as an Adjuvant for Lower Limb Nerve Blocks Following Oromaxillofacial Reconstruction
Brief Title: The Effect of Dexmedetomidine as an Adjuvant for Lower Limb Nerve Blocks
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaofeng Bai (Other)
Responsible Party: Sponsor-Investigator, Xiaofeng Bai, Associate Professor, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Dexmedetomidine in nerve block
Record Dates: First submitted 2017-03-16; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Free Flap Reconstruction
MeSH Terms: interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Placebo Comparator): Nerve blocks were administered with 0.3% ropivacaine without dexmedetomidine.
  Interventions: Drug: Ropivacaine
- Group RD (Experimental): Nerve blocks were administered with 0.3% ropivacaine and 50 μg dexmedetomidine.
  Interventions: Drug: 0.3% ropivacaine and 50 μg dexmedetomidine

INTERVENTIONS:
Drug: 0.3% ropivacaine and 50 μg dexmedetomidine — Nerve blocks were administered with 0.3% ropivacaine and 50 μg dexmedetomidine.
  Arms: Group RD
Drug: Ropivacaine — Nerve blocks were administered with 0.3% ropivacaine.
  Arms: Group R

SUMMARY:
Peripheral nerve block has been recommended as the technique for postoperative pain management because it provides equivalent analgesia but with fewer adverse effects than either systemic or epidural analgesia.

The use of clonidine, a partial α2 adrenoceptor agonist, has been reported to prolong the duration and analgesia in peripheral nerve blockade. Dexmedetomidine is a more selective and shorter-acting α2 adrenergic receptor.However, its use in femoral and common peroneal nerve blocks has not been described.

In this study, we investigated the effect of adding dexmedetomidine as additive in femoral and common peroneal nerve blocks for postoperative analgesia.

Patients, diagnosed as oromaxillofacial tumor and undergoing elective free fibular or anterolateral thigh flap reconstruction, were divided into two groups in a randomized, double-blind fashion. In Group Ropivacaine (Group R), nerve blocks were administered with 0.3% ropivacaine. In Group Ropivacaine + Dexmedetomidine (Group RD), nerve blocks were administered with 0.3% ropivacaine and 50 μg dexmedetomidine.The primary endpoints were the onset time and duration of sensory blocks. The secondary endpoints were heart rate, blood pressure, SpO2, sedation level, the duration of motor blocks.

DETAILED DESCRIPTION:
Peripheral nerve block has been recommended as the technique for postoperative pain management because it provides equivalent analgesia but with fewer adverse effects than either systemic or epidural analgesia.

The use of clonidine, a partial α2 adrenoceptor agonist, has been reported to prolong the duration and analgesia in peripheral nerve blockade. Dexmedetomidine is a more selective and shorter-acting α2 adrenergic receptor.However, its use in femoral and common peroneal nerve blocks has not been described.

In this study, we investigated the effect of adding dexmedetomidine as additive in femoral and common peroneal nerve blocks for postoperative analgesia.

Patients, diagnosed as oromaxillofacial tumor and undergoing elective free fibular or anterolateral thigh flap reconstruction, were divided into two groups in a randomized, double-blind fashion. For patients with free fibular flaps harvested, femoral nerve block and common peroneal nerve with ropivacaine were administered. For patients with anterolateral thigh flaps harvested, femoral nerve block with ropivacaine was administered.In Group R, nerve blocks were administered with 0.3% ropivacaine. In Group RD, nerve blocks were administered with 0.3% ropivacaine and 50 μg dexmedetomidine.The primary endpoints were the onset time and duration of sensory blocks. The secondary endpoints were heart rate, blood pressure, pulse oxygen saturation (SpO2), sedation level, the duration of motor blocks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of oral and maxillofacial tumor.
* Undergoing microsurgical oromandibular reconstruction with free fibular flaps or anterolateral thigh flaps.
* Greater than 18 years old.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* True allergy to local anesthetics or dexmedetomidine.
* History of chronic pain on opioids within the last 12 months.
* Specific mental health issues such as schizophrenia or bipolar disorder.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-20 (Estimated); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
the duration of sensory blocks | The duration of sensory blocks was recorded up to 48 hours after injection.
  The duration of sensory block was defined as the time interval between the end of ropivacaine administration and the pain score up to 5.

SECONDARY OUTCOMES:
sedation level | every 5 minutes until 30 minutes after injection, and then every 60 minutes up to 48 hours
  Sedation level was assessed using visual scale.
heart rate | every 5 minutes until 30 minutes after injection, and then every 60 minutes up to 48 hours
  If the heart rate is lower 50 beat/minute, atropine was administered.

CONTACTS AND LOCATIONS:
Locations (1):
- School & Hospital of Stomatology, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No